CLINICAL TRIAL: NCT01032733
Title: Biological Effects of Weight Loss Plus Exercise in Obese Older African-American Women: An Investigation of Aging-related Changes in Black and White Women
Brief Title: Biological Effects of Weight Loss In Older, Obese Women
Acronym: WL+E
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 3992006; P30AG028740 (NIH)
Record Dates: First submitted 2009-12-14; First posted 2009-12-15 (Estimated); Results first posted 2012-06-14 (Estimated); Last update posted 2012-06-14 (Estimated); Status verified 2012-05

CONDITIONS: Obesity; Sarcopenia
Keywords: Weight Loss; Physical Function; Oxidative Stress; Inflammation
MeSH Terms: conditions — Obesity; Sarcopenia; Weight Loss; Inflammation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lifestyle Counseling (Experimental): In the experimental condition, participants attended a group-based weight management session plus three supervised exercise sessions each week.
  Interventions: Behavioral: Lifestyle Counseling
- Educational Control (Placebo Comparator): Participants in the educational control group attended monthly health education lectures on topics unrelated to weight loss.
  Interventions: Other: Educational Control

INTERVENTIONS:
Behavioral: Lifestyle Counseling — In the WL+E group, participants attended a group-based weight management session plus three supervised exercise sessions each week.
  Other Names: Weight Loss plus Exercise Intervention
  Arms: Lifestyle Counseling
Other: Educational Control — Participants in the educational control group attended monthly health education lectures on topics unrelated to weight loss (e.g., skin protection).
  Other Names: Health Educational Group
  Arms: Educational Control

SUMMARY:
Obesity and sedentary lifestyle are associated with physical impairments and biological changes in older adults. Weight loss combined with exercise may reduce inflammation and may improve physical functioning in older adults who are overweight or obese and sedentary. However, the mechanisms by which weight change and exercise influence physical functioning and sarcopenia remain largely understudied. ions). In the WL+E group, participants attended a group-based weight management session plus three supervised exercise sessions each week throughout the entire study. During each exercise session, participants engaged in both aerobic activities (i.e., walking) and lower body resistance training of moderate intensity. The participants in the educational control group attended monthly health education lectures on topics relevant to older adults. It was hypothesized that participants assigned to the WL+E intervention would 1) lose a larger amount of weight, 2) improve their physical function levels, and 3) reduce levels of oxidative stress and inflammation to a greater degree than participants assigned to the Educational Control group. Outcomes are: 1) body weight, 2) walking speed (assessed by 400 meter walk test), 3) the Short Physical Performance Battery [SPPB], and 4) knee extension isokinetic strength. The objectives of this pilot study are fourfold: 1) to demonstrate the feasibility, acceptability, and efficacy of the proposed WL+E intervention in a sample of 40 sedentary, obese older adults with impaired physical functioning; 2) to examine the biological effects of the intervention on inflammatory processes, oxidative stress, apoptosis, sarcopenia, muscle and body composition, muscle strength, and functional performance; 3) to determine whether the expected beneficial effects of the WL+E intervention on physical functioning are mediated by changes in inflammation, apoptosis, and sarcopenia; and 4) to determine the effect size of the WL+E intervention on key outcomes and provide the basis for sample size calculations in the planning of a larger RCT.

DETAILED DESCRIPTION:
SPECIFIC AIMS A.1. Overview Obesity is associated with a higher level of inflammation and oxidative stress, which in turn are important mediators of sarcopenia, declines in physical functioning, and physical limitations in older adults. Several observational studies and randomized controlled trials (RCTs) suggest that behavioral interventions targeting weight loss through caloric restriction plus exercise (CR +EX) may reduce inflammation and may improve function in obese older adults.3 The mechanisms by which CR +EX may influence physical functioning and sarcopenia (the involuntary loss of skeletal muscle with age) remain largely understudied. It is proposed that CR +EX may avert sarcopenia by reducing inflammation, oxidative damage, and consequent apoptosis of skeletal muscle myocytes.

A.2. Objective of the Pilot Study

The proposed pilot study will lay the groundwork for a RCT of the effects of CR +EX on inflammation, oxidative stress, apoptosis, body composition, intramuscular fat, sarcopenia, muscle strength, and physical functioning in obese older adults. The specific objectives of the proposed study are as follows:

1. Demonstrate the feasibility, acceptability, and efficacy of the proposed intervention, including:

   1. Ability to recruit 40 sedentary, older obese adults with mild to moderate functional disability;
   2. High rate of attendance at treatment sessions (Mean > 75%); and
   3. Good response to treatment (Mean body weight loss > 7%).
2. Evaluate the biological effects of the CR +EX intervention, including changes in:

   1. Inflammation (i.e., tumor necrosis factor-α [TNF- α], interleukin-6 [IL-6], myeloperoxidase [MPO]);
   2. Oxidative stress (RNA and DNA oxidative damage in leucocytes)
   3. Apoptosis (as assessed by caspases and nuclear DNA fragmentation);
   4. Body composition (as assessed by dual x-ray absorptiometry [DXA)] and
   5. Sarcopenia and muscle composition (i.e., fat free muscle and intramuscular fat, as assessed by Magnetic Resonance Imaging [MRI] and Magnetic Resonance Spectroscopy [MRS]).
3. Examine functional changes associated with weight loss including:

   1. Upper and lower extremity muscle strength (as measured by grip strength and isometric and isokinetic ankle and knee strength);
   2. Response to the Short Physical Performance Battery; and
   3. Self-reported disability.
4. Test whether the expected beneficial effects of the CR +EX intervention on physical functioning are mediated by changes in inflammation, oxidative stress, apoptosis, and sarcopenia;
5. Determine the effect size of the CR +EX intervention on the key outcomes so as to provide the basis for sample size calculations for the planning of the larger RCT.

A.3. Research Hypotheses for the Future RCT

The synergistic effects of CR +EX may be effective in reversing the effects of inflammation, oxidative distress, apoptosis, and sarcopenia on both muscle strength and physical functioning in older adults. Thus, the primary goal of this pilot study is to provide support for a future RCT to test the hypothesis that a lifestyle intervention targeting a 7% loss in body weight through CR + EX will produce greater reductions in these outcomes, as compared to a (no weight loss) control condition. The future RCT would be designed to test the following primary and secondary hypotheses:

Primary hypotheses. As compared with a control condition, the CR +EX Intervention will:

1. Decrease inflammation (as measured by TNF-α, IL-6, and MPO);
2. Decrease oxidative stress (as measured by DNA and RNA damage in isolated leucocytes);
3. Decrease the rate of apoptosis (as measured by caspases and DNA laddering);
4. Produce favorable changes in body composition (i.e., a decrease in total fat mass and an increase in appendicular lean mass, as assessed by DXA); and
5. Produce favorable changes in muscle composition (i.e., a decrease in intramuscular fat and an increase in fat-free muscle as assessed by MRI/MRS).
6. Increase muscle strength and performance (as assessed through validated strength measures)

ELIGIBILITY:
Inclusion Criteria:

* African American or Caucasian Female
* Age between 55 - 79 years
* BMI > 28 kg/m2
* sedentary lifestyle (defined as < 20 min/week of aerobic exercise)
* mild to moderate physical impairments (score on the Short Physical
* Performance Battery between 4 - 10).

Exclusion Criteria:

* Weight >300 lbs.
* Weight loss > 10 lbs. within the past 6 months
* History of surgery for weight loss
* Hospitalization with the past 6 months
* Significant underlying disease likely to limit lifespan and/or increase risk of interventions (cancer or any condition with a life expectancy < 5 years with the exception of non-melanoma skin cancer; serious infectious diseases; myocardia infarction, cerebrovascular accident, or unstable angina within the past 6 months; NYHA Class 3 or 4 congestive heart failure; aortic stenosis; chronic hepatitis; cirrhosis; kidney disease; solid organ transplantation; chronic gastrointestinal disorders; fibromyalgia; chronic fatigue syndrome; major psychiatric disorder).
* Metabolic exclusions (resting blood pressure > 160/90 mmHg, fasting blood glucose > 160 mg/dl, fasting triglycerides > 400 mg/dl; patients on medication for hypertension, diabetes, or hyperlipidemia will not be excluded unless their values suggest "poor control").
* Medication exclusions (Antipsychotic agents; monoamine oxidase inhibitors; systemic corticosteroids; antibiotics for HIV or TB; chemotherapeutic drugs; or current use of prescription weight-loss drugs).
* Physical limitations likely to prevent exercise participation (use of walker; breathing problems that limit physical activity).
* Conditions or behaviors likely to affect the conduct of the trial (e.g., unwilling or unable to give informed consent; unwilling to accept random assignment; likely to move out of area within next 2 years; unable to attend weekly meetings; unwilling to complete paperwork; participation in another randomized research project; unwilling or unable to comply with study requirements or schedule)
* Contraindications to MRI (MR-incompatible implants or severe claustrophobia).
* Contraindications to muscle biopsy (i.e., lidocaine allergy)
* Presence of any other medical condition, which in the opinion of the research staff, would be incompatible with participation in the weight loss plus exercise program.

Ages: 55 Years to 79 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2006-09; Primary Completion 2009-08 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen D Anton, PhD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

REFERENCES:
- [Result] Anton SD, Manini TM, Milsom VA, Dubyak P, Cesari M, Cheng J, Daniels MJ, Marsiske M, Pahor M, Leeuwenburgh C, Perri MG. Effects of a weight loss plus exercise program on physical function in overweight, older women: a randomized controlled trial. Clin Interv Aging. 2011;6:141-9. doi: 10.2147/CIA.S17001. Epub 2011 Jun 15. PMID 21753869
- [Result] Wohlgemuth SE, Lees HA, Marzetti E, Manini TM, Aranda JM, Daniels MJ, Pahor M, Perri MG, Leeuwenburgh C, Anton SD. An exploratory analysis of the effects of a weight loss plus exercise program on cellular quality control mechanisms in older overweight women. Rejuvenation Res. 2011 Jun;14(3):315-24. doi: 10.1089/rej.2010.1132. Epub 2011 Jun 1. PMID 21631380

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited between September 2006 - December 2008 through a variety of methods including media articles, direct mailings, newspaper announcements, and presentations to community groups.
Pre-assignment Details: Following telephone screening, potentially eligible persons were invited to attend a screening visit during which the purposes and procedures of the study were explained and informed consent was obtained.
Period: Overall Study
Arm/Group | Lifestyle Counseling | Educational Control
Started | 17 | 17
Completed | 16 | 16
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lifestyle Counseling | Educational Control | Total
Number analyzed (Participants) | 17 | 17 | 34
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 11 | 23
  >=65 years | 5 | 6 | 11
Age Continuous [Mean (Standard Deviation); unit: years] | 63.7 (4.5) | 63.7 (6.7) | 63.7 (5.59)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 17 | 34
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 17 | 17 | 34

OUTCOME MEASURES:

1. Primary Outcome: Performance on the 400 Meter Walk
Description: Walking speed was assessed at baseline and 24-week assessment by the 400 Meter Walk Test, during which participants were asked to complete a standard walking course at their usual pace. Participants were permitted to stop during the walk but were not allowed to sit or receive help from others and were required to complete the course in 15 minutes.
Time Frame: 24 weeks
Population: Change from baseline (e.g., baseline and 24 weeks) was defined as the value at time t minus the value observed at baseline for all response measures. The five imputed responses sampled from a normal distribution with the mean baseline value (so 'centered' with a baseline carried forward mechanism).
Measure: Mean (Standard Deviation); unit: meters per second
Arm/Group | Lifestyle Counseling | Educational Control
Number analyzed (Participants) | 17 | 17
meters per second | 0.16 (0.03) | 0.02 (0.03)
Statistical Analysis 1: Comparison: Lifestyle Counseling vs Educational Control; This trial represented a pilot study, which was designed to demonstrate the feasibility, acceptability, and efficacy of the intervention; therefore, a power analysis was not conducted. The statistical analyses consisted of descriptive and intent-to-treat (ITT) modeling procedures; Test type: Superiority or Other; p < 0.05, ANCOVA; Median Difference (Net) = 0.06, Standard Deviation 0.5

2. Secondary Outcome: Body Weight
Description: Body weight was measured under fasting conditions following voiding in the morning at baseline and at the 24-week post-treatment assessment.
Time Frame: 24 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | Lifestyle Counseling | Educational Control
Number analyzed (Participants) | 17 | 17
kilograms | -5.95 (4.1) | -0.23 (4.08)
Statistical Analysis 1: Comparison: Lifestyle Counseling vs Educational Control; Test type: Superiority or Other; p < 0.05, ANCOVA; Mean Difference (Net) = 5, Standard Deviation 5

3. Secondary Outcome: Short Physical Performance Battery
Description: Scores on the Short Physical Performance Battery (SPPB) were obtained at baseline and at the 24-week post-treatment assessment visit. The SPPB consists of a 4 meter walk, repeated chair stands, and three hierarchical standing balance tests. The time to complete each of the three performance measures was assigned a categorical score based on normative data, ranging from 0 to 4. A summary score ranging from 0 (worst performers) to 12 (best performers) was calculated by adding walking speed, chair stands, and balance scores.
Time Frame: 24 weeks
Population: Change from baseline (e.g., baseline and 24 weeks) was defined as the value at time t minus the value observed at baseline for all response measures.
Measure: Mean (Standard Deviation); unit: score on the SPPB
Arm/Group | Lifestyle Counseling | Educational Control
Number analyzed (Participants) | 17 | 17
score on the SPPB | 1.82 (1.24) | 0.8 (1.20)
Statistical Analysis 1: Comparison: Lifestyle Counseling vs Educational Control; Test type: Superiority or Other; p < 0.05, Wilcoxon (Mann-Whitney); Mean Difference (Net) = 2, Standard Deviation 2

4. Secondary Outcome: Knee Extension Maximum Isokinetic Strength (Weight Lifted in Kilograms).
Description: Maximal knee extension strength using each participant's strongest leg was measured using a Biodex. The participants were asked to develop their maximal isokinetic knee extension strength. Three trials of 5 repetitions were performed and the peak torque value was used for statistical analyses.
Time Frame: 24 weeks
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | Lifestyle Counseling | Educational Control
Number analyzed (Participants) | 17 | 17
kilograms | 4.33 (14.35) | 3.95 (14.43)
Statistical Analysis 1: Comparison: Lifestyle Counseling vs Educational Control; Test type: Superiority or Other; p < 0.05, ANCOVA; Mean Difference (Net) = 5, Standard Deviation 15

5. Secondary Outcome: Mitochondrial Function (Cox IV Subunit)
Description: Western blot analysis was performed to determine complex content. The amount of Cox IV subunit was determined for each Reporting Group via Western Blot analysis at baseline and week 24.
Time Frame: 24 weeks
Population: Change from baseline (e.g., baseline and 24 weeks) was defined as the value at time t minus the value observed at baseline for all response measures. In addition, the discrepancy for the number of participants is becasue we could only obtain information on a subset of participants due to the nature of the procedure (muscule biopsy).
Measure: Mean (Standard Deviation); unit: fold change (ug/ml)
Arm/Group | Lifestyle Counseling | Educational Control
Number analyzed (Participants) | 5 | 7
fold change (ug/ml) | 1.65 (0.59) | 1.21 (0.31)
Statistical Analysis 1: Comparison: Lifestyle Counseling vs Educational Control; Test type: Superiority or Other; p < 0.05, Wilcoxon (Mann-Whitney); Mean Difference (Net) = 1, Standard Deviation 1

ADVERSE EVENTS:
Time Frame: Adverse events were assessed between baseline and six months.
Arm/Group | Lifestyle Counseling | Educational Control
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/17
Other Adverse Events (participants affected / at risk) | 7/17 | 5/17
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lifestyle Counseling (N=17) | Educational Control (N=17)
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 7 (7) | 5 (5)

LIMITATIONS AND CAVEATS:
Limitations include the following: (1) the sample size was relatively small,(2)the study was not adequately powered to detect differences between African American and Caucasian women in response to the intervention, (3) inclusion of only women.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No